CLINICAL TRIAL: NCT05055843
Title: Novel Synthetic T2W MR Imaging and Spin Parameter Mapping Techniques for Prostate Cancer Without an Endorectal Coil
Brief Title: Novel Synthetic T2W MR Imaging and Spin Parameter Mapping Techniques for Screening Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2021-0273; NCI-2021-05282 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0273 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-07-21; First posted 2021-09-24 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Prostate Adenocarcinoma; Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (3D MRI) (Experimental): Patients undergo 3D MRI imaging over 15 minutes with standard of care MRI or at a separate time.
  Interventions: Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging — Undergo 3D MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This clinical trial studies examines a 3D magnetic resonance imaging (MRI) compared to standard MRI imaging techniques in screening patients with prostate cancer. Diagnostic procedures, such as MRI, may help find and diagnose prostate cancer. Computer systems that allow doctors to create a 3-dimensional (3-D) picture of the tumor may help in planning.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether the image quality of the novel 3-dimensional (3D) T2-weighted imaging (T2W) synthetic imaging technique without endorectal coil is comparable to the 2-dimensional (2D) T2W imaging technique without endorectal coil.

SECONDARY OBJECTIVE:

I. To evaluate the qualitative diagnostic quality of the T2W images provided by the novel 3D technique, as determined by subjective scoring by experienced readers.

EXPLORATORY OBJECTIVE:

I. To investigate the feasibility of novel 3D synthetic imaging and multi-spin parameter mapping technique of prostate for the detection of clinically significant prostate cancer (csPCa).

OUTLINE:

Patients undergo 3D MRI imaging over 15 minutes with standard of care MRI or at a separate time.

ELIGIBILITY:
Inclusion Criteria:

* Male, age >= 18
* Untreated, biopsy-proven with intermediate and high-risk adenocarcinoma of the prostate
* Patient is being considered for curative-intent treatment with radical prostatectomy
* Patient has provided written informed consent for participation in this trial
* Patient should be eligible for scanning on a 3T magnet

Exclusion Criteria:

* Low-risk adenocarcinoma of prostate
* Any prior therapy for prostate cancer
* A history of other active malignancy within the last 2 years
* Prostate cancer with significant sarcomatoid, spindle cell, or neuroendocrine small cell components
* Cardiac pacemaker
* Orthopedic hardware in the pelvis and spine
* Claustrophobia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
To be assessed with scoring of quantitative image metrics in regions of prostate cancer and benign tissue | through study completion, an average of 1 year
  Comparing the 2-dimensional (2D) T2W imaging technique without endorectal coil.
  Scored from 1 to 5 with PI-RADS 1 indicating that csPCa is highly unlikely whereas a PI-RADS 5 score indicates that csPCa is highly likely to be present.

CONTACTS AND LOCATIONS:
Overall Officials: Tharakeswara Bathala, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org